CLINICAL TRIAL: NCT05689411
Title: The Effect of The Musical Toy Used During Peripheral Vascular Access on Children's Pain, Fear And Parents' Satisfaction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ordu University (Other)
Responsible Party: Principal Investigator, Dilek Kucuk Alemdar, Associate professor, Ordu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: KAEK291
Record Dates: First submitted 2022-12-29; First posted 2023-01-19 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Pain; Child, Only; Parents
Keywords: Pain; Fear; Children; Parent
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: randomized controlled experimental
Who Masked: Outcomes Assessor
Masking Description: the database of the research will be created by a university graduate statistician working in a statistical center independent of the research, apart from the researcher.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Musical Toy Group (Experimental): The child and his parents in the experimental group were distracted by playing with the xylophone, a musical toy, 5 minutes before the peripheral vascular access procedure. The xylophone is a percussion wooden toy. There are two wooden bars on the xylophone that make melodious sounds when the metal plates are struck. The xylophone toy was introduced to the child and the parent, and they were given the opportunity to examine it. Before the procedure, one of the wooden sticks of the toy was given to the child and the other to the parent. Before, during and after the procedure, the child and his parents played together by making a melodic sound from the musical toy xylophone. While the child and his parents were playing with the toy, the researcher attached a tourniquet to the appropriate extremity of the child and determined the vein to which the vascular access would be performed.
  Interventions: Device: Musical Toy
- Control Group (No Intervention): No distraction technique was applied to the children in the control group before the vascular access procedure. After the procedure was explained according to the child's developmental level, the researcher applied the procedure to open a vascular access in accordance with the institutional policies.

INTERVENTIONS:
Device: Musical Toy — The child and his parents in the experimental group were distracted by playing with the xylophone, a musical toy, 5 minutes before the peripheral vascular access procedure. The xylophone is a percussion wooden toy. There are two wooden bars on the xylophone that make melodious sounds when the metal plates are struck. The xylophone toy was introduced to the child and the parent, and they were given the opportunity to examine it. Before the procedure, one of the wooden sticks of the toy was given to the child and the other to the parent. Before, during and after the procedure, the child and his parents played together by making a melodic sound from the musical toy xylophone. While the child and his parents were playing with the toy, the researcher attached a tourniquet to the appropriate extremity of the child and determined the vein to which the vascular access would be performed.
  Arms: Musical Toy Group

SUMMARY:
The research was carried out as a randomized controlled experimental study in order to examine the effects of the child's pain, fear and parent's satisfaction before and after vascular access with a musical toy-xylophone, which is used as a distraction technique for the preparation of the 3-6 year old child hospitalized in the pediatric clinic.

DETAILED DESCRIPTION:
The population of the study consists of children aged 3-6 years who applied to Durağan Şehit Hakan Tanrıkulu State Hospital Pediatric Service between January 2022 and December 2022 and needed vascular access. The sample of the study consisted of 70 children (control: 35, experiment: 35) who met the case selection criteria. Child and Parent Descriptive Information Form, Child Fear Scale (CFS), Children's Emotional Indicator Scale (CEIS), QUCHER Photographic and Numerical Rating Form (QUCHER), and Nurse-Patient Collaboration Level and Parent Satisfaction Form were used. While the children in the experimental group were playing with a musical toy with their parents, peripheral vascular access was performed.

ELIGIBILITY:
Inclusion Criteria:

* The child is between 3-6 years old,
* Volunteering of parents and children to participate in the research,
* The child does not come to the hospital with acute pain,

Exclusion Criteria:

* The child has a hearing, vision and mental problem,
* The child and the parent do not understand and speak Turkish easily,
* Absence of a primary caregiver,

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Children's Emotional Indicator Scale | 5 minutes before the procedure.
  children's emotional behaviors during stressful medical procedures.It takes a value between 1 and 5 for each category. The total score that can be obtained from the scale varies between 5-25. As the scores obtained from the scale increase, negative emotional indicators increase.
Children's Emotional Indicator Scale | 5 minutes after the procedure.
  children's emotional behaviors during stressful medical procedures.It takes a value between 1 and 5 for each category. The total score that can be obtained from the scale varies between 5-25. As the scores obtained from the scale increase, negative emotional indicators increase.
Child Fear Scale | 5 minutes before and after the procedure.
  The CFS consists of five drawn facial expressions ranging from a neutral expressioanxiety level of children.The mean score of the CFS is 1.9 ± 0.1 (min=0, max=4). The CLS can also be scored by the parent and the researcher.
Child Fear Scale | 5 minutes before the procedure.
  The CFS consists of five drawn facial expressions ranging from a neutral expressioanxiety level of children.The mean score of the CFS is 1.9 ± 0.1 (min=0, max=4). The CLS can also be scored by the parent and the researcher.
  anxiety level of children.
Qucher-Photographic and Numerical Rating Scale | 5 minutes before the procedure.
  The Qucher scale can be used in children aged 3-12 years.Pain intensity is evaluated from 0 as "pain-no pain" and up to 10 as "the greatest pain-pain you can have".
Qucher-Photographic and Numerical Rating Scale | 5 minutes after the procedure.
  The Qucher scale can be used in children aged 3-12 years.Pain intensity is evaluated from 0 as "pain-no pain" and up to 10 as "the greatest pain-pain you can have".

SECONDARY OUTCOMES:
Nurse-Patient Cooperation and Patient Parent Satisfaction Form | 5 minutes before the procedure.
  The Nurse-Patient Collaboration section consists. The patient is asked to rate how his or her compliance with the procedure is between 0 and 10 points. 0 represents the worst fit and 10 the best fit.questions directed to the nurse performing the procedure.
Nurse-Patient Cooperation and Patient Parent Satisfaction Form | 5 minutes after the procedure.
  The Nurse-Patient Collaboration section consists. The patient is asked to rate how his or her compliance with the procedure is between 0 and 10 points. 0 represents the worst fit and 10 the best fit.questions directed to the nurse performing the procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- Dilek alemdar, Ordu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No